CLINICAL TRIAL: NCT06415331
Title: Comparison of The Effectiveness Between Conventional Therapy and Conventional Therapy Plus Pulsed-Radiofrequency in Herniated Nucleus Pulposus Patients at Dr. Saiful Anwar Hospital, Malang
Brief Title: Effectiveness of Conventional Therapy Plus Pulsed-Radiofrequency for Herniated Nucleus Pulposus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Syaiful Anwar Hospital, Malang (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSSA-00124
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Herniated Nucleus Pulposus; Pain
MeSH Terms: conditions — Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Subjects in this arm received interventions which were conventional, including opioid and non-opioid analgesics, adjuvant analgesics, muscle relaxants, and physiotherapy.
  Interventions: Other: Conventional therapy
- Conventional therapy + pulsed radiofrequency (Experimental): Subjects in this arm received pulsed radiofrequency in addition to the same conventional therapy as the other arm.
  Interventions: Procedure: Pulsed radiofrequency; Other: Conventional therapy

INTERVENTIONS:
Procedure: Pulsed radiofrequency — Individualized dose of pulsed radiofrequency is given for 6 minutes.
  Arms: Conventional therapy + pulsed radiofrequency
Other: Conventional therapy — Conventional therapy for HNP consisting of:
  * Acetaminophen
  * NSAID: Etoricoxib, celecoxib, meloxicam, diclofenac, ibuprofen
  * Muscle relaxant: eperisone, diazepam
  * Opioid: codein, tramadol
  * Adjuvant analgesics: Amitriptyline, pregabalin, gabapentin
  * Physiotherapy: Short wave diathermy, ultrasound diathermy, transcutaneous electrical nerve stimulation, and exercise

SUMMARY:
The purpose of this research was to study whether the additional application of a certain medical intervention making use of radiofrequencies (pulsed-radiofrequency) would reduce pain in patients with herniated disk.

DETAILED DESCRIPTION:
Pain is an uncomfortable sensory and emotional experience that can affect quality of life. Low back pain (LBP) is one of the most common causes of pain, with herniated nucleus pulposus (HNP) being a common etiology. Pulsed radiofrequency (PRF) is a relatively novel technique that has shown promising results in many applications, including spinal pain conditions.

This quasi-experimental study aimed to compare pain levels between patients who underwent conventional therapy (CT) alone and CT plus PRF as management in patients with HNP. Pain severity was measured in the numeric rating scale before and 1 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having an established diagnosis of HNP
* Complaint present for at least the pas 3 months
* Experiencing pain intensity of 4 or greater on the numeric rating scale
* Capable of giving informed consent

Exclusion Criteria:

* Pregnant patients
* Presence of infection at the site of pulsed radiofrequency
* HNP with red flags.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
Pain severity | 1 month after treatment
  Pain severity measured with the numeric rating scale (NRS). The numeric rating scale measures pain on a scale of 0-10 with 0 representing "no pain" and 10 representing "the worst pain possible".

CONTACTS AND LOCATIONS:
Overall Officials: Hana H Fachir, M.D., Principal Investigator — Faculty of Medicine, Universitas Brawijaya, Malang, Indonesia
Locations (1):
- Dr. Saiful Anwar Hospital, Malang, East Java, Indonesia